CLINICAL TRIAL: NCT04222309
Title: Laparoscopically Harvested Omental Free Tissue Autograft to Bypass the Blood Brain Barrier (BBB) in Human Recurrent Glioblastoma Multiforme (rGBM)
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Per IRB closed and opened a new study.
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, John Boockvar, MD Zucker SOM @Hofstra/Northwell, Principal Investigator, Northwell Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-0801
Record Dates: First submitted 2020-01-06; First posted 2020-01-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Glioma; Glioma, Malignant; Glioblastoma; Glioblastoma Multiforme; Glioblastoma Multiforme of Brain; GBM; Brain Cancer
Keywords: blood brain barrier; omental free flap
MeSH Terms: conditions — Glioma; Glioblastoma; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Laparoscopically harvested omental free flap (Experimental): 1. Standard neurosurgical removal of recurrent GBM,
  2. Removal of fat from the abdomen called omentum using a camera (laparoscopically),
  3. Lining the brain tumor cavity with the piece of omentum,
  4. Joining the blood vessels of the omentum to blood vessels in the scalp or neck to ensure that it maintains good blood flow.
  Interventions: Procedure: Laparoscopically harvested omental free flap

INTERVENTIONS:
Procedure: Laparoscopically harvested omental free flap — Laparoscopically harvested omental free flap into the resection cavity of recurrent glioblastoma multiforme (GBM) patients.

SUMMARY:
This single center, single arm, open-label, phase I study will assess the safety of a laparoscopically harvested omental free flap into the resection cavity of recurrent glioblastoma multiforme (GBM) patients.

All participants included in the study will undergo standard surgical resection for diagnosed recurrent GBM. Following the resection, the surgical cavity will be lined with a laparoscopically harvested omental free flap. The participant's dura, bone and scalp will be closed as is customary. The participant will be followed for side effects within 72 hours, 7 days, 30 days, 90 days and 180 days. Risk assessment will include seizure, stroke, infection, tumor progression, and death.

DETAILED DESCRIPTION:
Laparoscopically harvested omental free flaps are commonly used to fill surgical cavities after resection of head and neck cancers. The investigators hypothesize that a laparoscopically harvested omental free flap in our patients with resected recurrent GBM may be used as a readily available and accessible means of circumventing the blood brain barrier (BBB) selectively and focally. The laparoscopically harvested omental free flap with its long vascular pedicle length, wide rotational arc and available surface area would easily conform to many resected GBM cavities in our human patients with acceptable risk. The predictable and rich vascular anatomy of a laparoscopically harvested omental free makes it an ideal flap for cases of previously irradiated and/or infected wound beds. This is why it is successfully used in head and neck and skull base tumors. The permeability of the blood vessels of the laparoscopically harvested omental free flap should allow for improved delivery of chemotherapeutics and immune cells (macrophages and T cells) into the vicinity, extracellular space and microenvironment of the resected tumor cavity including the brain adjacent to the tumor (BAT). "Milky spots" within the omentum will also provide direct deposition of immune cells such as dendritic, macrophages and lymphocytes into the milieu of the resected GBM.

The investigators aim to prove that this commonly surgical technique for head and neck cancers is safe in a small human cohort of patients with resected recurrent GBM and may improve progression-free survival (PFS).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a male or female 18 years of age or older.
2. Subject is undergoing planned resection of known or suspected GBM.
3. Subject has a Karnofsky Performance Status (KPS) 70% or greater.
4. Subject has a life expectancy of at least 6 months, in the opinion of the Investigator.
5. Based on the pre-operative evaluation by neurosurgeon, the subject is a candidate for ≥ 80% resection of enhancing region.
6. Subject must be able to undergo MRI evaluation.
7. Subject meets the following laboratory criteria:

   1. White blood count ≥ 3,000/µL
   2. Absolute neutrophil count ≥ 1,500/µL
   3. Platelets ≥ 100,000/µL
   4. Hemoglobin > 10.0 g/dL (transfusion and/or ESA allowed)
   5. Total bilirubin and alkaline phosphatase ≤ 2x institutional upper limit of normal (ULN)
   6. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3 x ULN
   7. Blood urea nitrogen (BUN) and creatinine < 1.5 x ULN
8. Females of reproductive potential must have a negative serum pregnancy test and be willing to use an acceptable method of birth control.
9. Able to understand and willing to sign an institutional review board (IRB)-approved written informed consent document

Inclusion criteria considered during surgery:

1. Subject has a histologically confirmed (frozen section) diagnosis of recurrent WHO Grade IV glioblastoma multiforme (GBM).
2. Omental free flap is technically feasible.

Exclusion Criteria:

1. Subject, if female, is pregnant or is breast feeding.
2. Subject intends to participate in another clinical trial.
3. Subject intends to undergo treatment with the Gliadel® wafer at the time of this surgery.
4. Subject has an active infection requiring treatment.
5. Subject has radiographic evidence of multi-focal disease or leptomeningeal dissemination.
6. Subject has a history of other malignancy, unless the patient has been disease-free for at least 5 years. Adequately treated basal cell carcinoma or squamous cell skin cancer is acceptable regardless of time, as well as localized prostate carcinoma or cervical carcinoma in situ after curative treatment
7. Subject has a known positive test for human immunodeficiency virus infection, or active hepatitis B or hepatitis C infection.
8. Subject has a history or evidence of any other clinically significant disorder, condition or disease that would pose a risk to subject safety or interfere with the study evaluation, procedures or completion.
9. Subject has had prior abdominal surgery.
10. Subject has severe renal insufficiency rendering gadolinium MRI contraindicated.
11. Subject who are unable to have an MRI scan for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-01-06 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Safety parameter: proportion of patients experiencing rapidly progressive disease as indicated by MRI using RANO Criteria | Study Day 1-180
  Increase in tumor size relative to baseline will be measured using RANO and assessed by MRI throughout study at within 72 hours, 7 days, 30 days, 90 days and 180 days. Rapidly progressive disease is defined as 25% growth relative to baseline.
Safety parameter: proportion of patients experiencing increase in seizures, stroke, and infection | Time Frame: Study Day 1-180
  Increase in seizures (defined as 15% relative to baseline), occurrence of a stroke, or occurrence of a severe infection will be determined throughout study within 72 hours, 7 days, 30 days, 90 days and 180 days.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 6 months
  The proportion of patients who are alive at 6 months from flap implantation and are progression-free will be estimated using standard methods for proportions, along with the associated exact 95% confidence interval.
Overall Survival (OS) | 6 months
  OS will be calculated as the time from treatment initiation (flap implantation) to the time of death.
Percent of screen fails | Study Day 1 - 24 months
  The number and percent of screen failures with the reason for screen failures (flap not viable etc.) will be tabulated and summarized.

CONTACTS AND LOCATIONS:
Overall Officials: John Boockvar, MD, Principal Investigator — Northwell Health
Locations (1):
- Lenox Hill Brain Tumor Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No